CLINICAL TRIAL: NCT01130753
Title: A Phase II Trial of Neoadjuvant Erlotinib (Tarceva®) Followed by Surgery for Selected Patients With Stage IIIA, N2-positive Non-Small Cell Lung Cancer
Brief Title: Efficacy of Erlotinib in Neoadjuvant Setting in Patients With Stage IIIA, N2-positive Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Keunchil Park, Principal investigator, Samsung Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-08-029
Record Dates: First submitted 2010-05-17; First posted 2010-05-26 (Estimated); Last update posted 2013-05-30 (Estimated); Status verified 2013-05

CONDITIONS: Lung Neoplasms; Erlotinib; Neoadjuvant Therapy
MeSH Terms: conditions — Lung Neoplasms | interventions — Erlotinib Hydrochloride

INTERVENTIONS:
Drug: Erlotinib — Erlotinib 150mg per day for 8 weeks

SUMMARY:
This study propose neoadjuvant chemotherapeutic role by erlotinib.

DETAILED DESCRIPTION:
It is widely accepted that patients with locally advanced non-small cell lung cancer would have better outcome with neoadjuvant therapy followed by surgery than surgery alone. However what should be the standard treatment option is still unclear.

Erlotinib (Tarceva®)is an oral inhibitor of epidermal growth factor receptor (EGFR) tyrosine kinase and its anti-neoplastic effect is approved especially women, patients with adenocarcinoma, non-smoker and Asian population. Moreover if the malignant tissue has EGFR mutation, its efficacy is known to be enhanced.

So we expect that in those population, patients with locally advanced, N2 positive, erlotinib would be more beneficial than conventional cytotoxic chemotherapy in safety and convenience as neoadjuvant therapy.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed N2 positive and stage IIIA non-small cell lung cancer
* Has more than 2 conditions out of following 3 conditions ; adenocarcinoma, non-smoker, women
* Age ≥ 18 years and ECOG performance 0~1
* Has measurable lesion by RECIST 1.1
* No previous chemotherapy or radiation therapy
* Adequate organ function by following; ANC ≥1,500/uL, hemoglobin ≥9.0g/dL, platelet ≥100,000/uL, PaO2 ≥ 60 mmHg, Serum Cr < 1 x UNL or creatinine clearance > 60 ml/min, Serum bilirubin < 1 x UNL, AST (SGOT) and ALT (SGPT) < 2.5 x UNL, alkaline phosphatase < 5 x UNL
* Written informed consent form

Exclusion Criteria:

* Pulmonary carcinoid tumor
* Previous chemotherapy or radiation therapy
* Previous history of malignancy within 5 years from study entry except treated non-melanomatous skin cancer or uterine cervical cancer in situ
* Known allergic history of erlotinib
* Interstitial lung disease or fibrosis on chest radiogram
* Active infection, uncontrolled systemic disease (cardiopulmonary insufficiency, fatal arrhythmias, hepatitis)
* Pregnant or nursing women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2007-01; Primary Completion 2010-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Pathologic down-staging | 36 months

SECONDARY OUTCOMES:
Response rate | 36 months
Toxicity | 36 months
Progression free survival | 36 months
Overall survival | 36 months

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea